CLINICAL TRIAL: NCT00641875
Title: The Effect of Nocturnal Haemodialysis on Arterial Stiffness
Status: Completed | Type: Observational
Sponsor: Melbourne Health (Other)
Responsible Party: Sponsor
Other Study IDs: 2004.050
Record Dates: First submitted 2008-03-17; First posted 2008-03-24 (Estimated); Last update posted 2015-04-27 (Estimated); Status verified 2015-04

CONDITIONS: End Stage Renal Disease; Arterial Stiffness
Keywords: arterial stiffness; artery; aortic pulse wave velocity; pulse wave analysis; augmentation index; end stage renal disease; nocturnal hemodialysis; extended hours of hemodialysis; cardiovascular; hemodialysis
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Nocturnal Hemodialysis

SUMMARY:
Arterial stiffness refers to the accumulation of extracellular deposits of matrix and calcium which reduce blood vessel compliance. Although there is growing evidence that increased arterial stiffness is associated with chronic kidney disease (CKD), its pathogenesis is unclear. Pulse wave velocity (PWV) and augmentation index (AIx) provide tools for estimating arterial stiffness, and therefore predicting cardiovascular morbidity and mortality. The aims of the study are: (1) compare the effects of nocturnal and conventional haemodialysis on arterial stiffness, and (2) examine the relationship between arterial stiffness and clinical and biochemical parameters.

ELIGIBILITY:
Inclusion Criteria:

* adult dialysis patients
* able to perform home nocturnal haemodialysis

Exclusion Criteria:

* age < 18 and > 80 years
* any patient who is anticipating a live renal transplantation in forthcoming 12 months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All participants are adult patients who are receiving maintenance dialysis at the North West Dialysis Service. Consecutive patients enrolled in the Nocturnal Haemodialysis program are invited to participate in the study
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2005-12; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
To purpose of this study is to evaluate the arterial stiffness in subjects who have undergone 12 months nocturnal haemodialysis. | 12 months

SECONDARY OUTCOMES:
To examine the relationship between arterial stiffness and clinical and biochemical parameters | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael Lian, FRACP, MBBS, Principal Investigator — Department of Nephrology, Melbourne Health